CLINICAL TRIAL: NCT06027151
Title: Comparing the Efficacy of Metronidazole and Minocycline Gels for the Treatment of Diabetic Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/IIMC/IRC/22/2070
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis; Diabetes Mellitus
Keywords: Chronic periodontitis; Minocycline gel; Scaling and root planning; Metronidazole gel; Efficacy of local administration; Diabetes mellitus
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus; Chronic Periodontitis | interventions — Metronidazole; Minocycline

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind, patient was unaware of which drug they were administered. It was done by covering the syringes with colored tapes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Scaling and root planning (No Intervention): Once the patients fulfill the inclusion criteria and are randomly assigned to this group, they undergo scaling and root planning by the consultant. Baseline values are recorded, and patients are advised oral hygiene instructions i.e., proper brushing and flossing. They are recalled after 7 and 15 days and all clinical parameters are rerecorded.
- Scaling and root planning plus metronidazole gel (Experimental): After fulfilling the inclusion criteria and randomly assigning to this group, they undergo scaling and root planning by the consultant. Baseline values are recorded, and 1ml of 1% metronidazole gel is applied subgingivally. The patients are instructed not to spit or rinse for at least one hour. Then patients are advised oral hygiene instructions i.e., proper brushing and flossing. They are recalled after 7 and 15 days and all clinical parameters are rerecorded.
  Interventions: Drug: 1ml of 1% metronidazole gel
- Scaling and root planning plus minocycline gel (Experimental): After fulfilling the inclusion criteria and being randomly assigned to this group, the patients undergo scaling and root planning by the consultant. Baseline values are recorded, and 1ml of 2% minocycline gel is applied subgingivally. The patients are instructed not to spit or rinse for at least one hour. Then patients are advised oral hygiene instructions i.e., proper brushing and flossing. They are recalled after 7 and 15 days and all clinical parameters are rerecorded.
  Interventions: Drug: 1ml of 2% minocycline gel
- Scaling and root planning plus combination of metronidazole and minocycline gels (Experimental): After fulfilling the inclusion criteria and being randomly assigned to this group, the patients undergo scaling and root planning by the consultant. Baseline values are recorded, 1ml of the combination of 1% metronidazole gel and 2% minocycline gel is applied subgingivally. The patients are instructed not to spit or rinse for at least one hour. Then patients are advised oral hygiene instructions i.e., proper brushing and flossing. They are recalled after 7 and 15 days and all clinical parameters are rerecorded.
  Interventions: Drug: 1ml of combination of 1% metronidazole gel and 2% minocycline

INTERVENTIONS:
Drug: 1ml of 1% metronidazole gel — Subgingivally at baseline visit
  Other Names: metronidazole
  Arms: Scaling and root planning plus metronidazole gel
Drug: 1ml of 2% minocycline gel — sub gingivally at baseline visit
  Other Names: minocycline
  Arms: Scaling and root planning plus minocycline gel
Drug: 1ml of combination of 1% metronidazole gel and 2% minocycline — subgingivally at baseline visit
  Other Names: metronidazole/minocycline
  Arms: Scaling and root planning plus combination of metronidazole and minocycline gels

SUMMARY:
This clinical study randomized 380 diabetic chronic periodontitis patients into 4 groups: scaling and root planning alone (group I), scaling and root planning plus metronidazole gel (group II), scaling and root planning plus minocycline gel (group III), and scaling and root planning plus both metronidazole and minocycline gels (group IV). Periodontal measurements including probing depth, gingival color and texture, bleeding on probing, clinical attachment level, and recession were recorded at baseline, 7 days, and 15 days.

DETAILED DESCRIPTION:
It was a clinical trial with four arms. The research was carried out at the Pharmacology Department, IIMC Riphah University, Rawalpindi. The sample size was calculated to be 380 using the prevalence of disease, z-score, and 5% margin of error. Written informed consent was obtained from the participants. The patients being treated for chronic periodontitis were randomly divided into four groups (I, II, III, and IV). Patients in Group I were subjected to Scaling and root planning alone. Group II patients were given metronidazole gel following Scaling and root planning. Minocycline gel was locally applied subsequent to scaling and root planning in Group III patients. The combination of metronidazole gel and minocycline gel was administered after Scaling and root planning in Group IV patients. Scaling and root planning of all the patients was done. Periodontal probing depth, the color of the gingiva, texture of the gingiva, bleeding on probing, clinical attachment level, and recession were recorded for each patient at baseline visit, after 7 days, and after 15 days to determine and compare the efficacy of local administration of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed diabetic patients on either hypoglycemics or insulin therapy suffering from periodontitis

Exclusion Criteria:

Pregnant or nursing mothers Patients with gestational diabetes Alcoholics Patients under any anti-inflammatory or antibiotic drugs (daily for ˃7 consecutive days) within the last two months of elimination before entering the study.

Known allergy to minocycline, or metronidazole. Periodontal surgeries in the past Smoking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
PERIODONTAL POCKET DEPTH (PPD) | 15 days
  Periodontal pocket depth was measured in mm using a WHO (CPITN) periodontal probe.
  Baseline periodontal probing depth was measured before application of drug. It was remeasured on 7th day and 15th day. Reduction in probing depth indicates improvement on follow up visits.

SECONDARY OUTCOMES:
COLOR OF GINGIVA | 15 days
  Color of gingiva is observed at baseline visit, on 7th day and 15th day. Healthy gingiva is coral pink in color while diseased gingiva is erythematous cyanotic.
TEXTURE OF GINGIVA | 15 days
  Texture of gingiva is observed at baseline visit, on 7th day and 15th day. Healthy gingiva is matte and stippled. Diseased gingiva is smooth and shiny.
BLEEDING ON PROBING (BOP) | 15 days
  It was determined whether the site was bleeding on probing or not. Bleeding on probing is observed on the baseline visit, 7th day, and 15th day. If the gingiva is not bleeding then it is considered as normal.
CLINICAL ATTACHMENT Level | 15 days
  Distance from cementoenamel junction to depth of pocket is measured with the help of CPITN probe. Readings are taken on baseline visit, 7th day and 15th day. Severity index is as follows.
  Healthy gingiva- 0mm CAL Mild: 1- or 2-mm CAL Moderate: 3- or 4-mm CAL Severe: ≥ 5mm CAL
RECESIION OF GINGIVAL MARGIN: | 15 days
  Recession is measured from CEJ to margin of gingiva with the help of CPITN probe on baseline visit, 7th day and 15th day. Severity of disease is assessed as follows
  CLASS I:
  Marginal tissue recession that does not extend to the mucogingival junction. There is no loss of bone or soft tissue in the interdental area. This can be narrow or wide.
  CLASS II:
  Marginal tissue recession that extends to or beyond the mucogingival junction. There is no loss of bone or soft tissue in the interdental area. This can be narrow or wide.
  CLASS III:
  Marginal tissue recession that extends to or beyond the mucogingival junction. In addition, there is loss of bone and/or soft tissue in the interdental area or there is malpositioning of the tooth.
  CLASS IV:
  Marginal tissue recession that extends to or beyond the mucogingival junction with severe loss of bone and soft tissue interdentally and/or severe malpositioning of the tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Aeman Choudhary, BDS, Principal Investigator — Riphah International University, Rawalpindi
Locations (1):
- Islamic International Medical Collège, IIMC, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No